CLINICAL TRIAL: NCT05126342
Title: A Pilot Study to Estimate Efficacy of Combining Dostarlimab and Niraparib in Patients With Relapsed EOC After Treatment With PARPi
Brief Title: Study to Estimate Efficacy of Combining Dostarlimab and Niraparib in Relapsed EOC After Treatment With PARPi
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has been withdrawn; was never submitted to Competent authority nor to ethics commitee.
Sponsor: AGO Research GmbH (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OVAR 2.35; 2021-003572-14 (EudraCT Number)
Record Dates: First submitted 2021-10-18; First posted 2021-11-19 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Ovarian Cancer; Recurrent Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: Recurrent Ovarian Cancer; Niraparib; Dostarlimab
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — niraparib; dostarlimab

STUDY DESIGN:
Intervention Model Description: The study population will be divided into 2 cohorts:
  Cohort A: Recurrent ovarian-, fallopian tube, or primary peritoneal cancer with relapse after more than 6 months of PARPi maintenance therapy.
  Cohort B: Recurrent ovarian-, fallopian tube, or primary peritoneal cancer with relapse within 6 months of PARPi mainte-nance therapy.
  Both cohorts will receive the selective PARP 1/2 inhibitor niraparib in combination with the anti-PD-1 checkpoint inhibitor dostarlimab (TSR-042).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Recurrent ovarian-, fallopian tube, or primary peritoneal cancer with relapse after more than 6 months of PARPi maintenance therapy.
  Interventions: Drug: Niraparib; Drug: Dostarlimab
- Cohort B (Experimental): Recurrent ovarian-, fallopian tube, or primary peritoneal cancer with relapse within 6 months of PARPi maintenance therapy.
  Interventions: Drug: Niraparib; Drug: Dostarlimab

INTERVENTIONS:
Drug: Niraparib — Niraparib starting dose of study treatment will be based upon the patient's baseline body weight and baseline platelet count. Patients with a baseline body weight ≥77 kg and baseline platelet count ≥150 x 10^9/L may start with niraparib 300 mg (3 x 100 mg capsules) daily unless the dose has not already been reduced to 200 mg in a prior treatment line. Patients with a baseline body weight <77 kg or a baseline platelet count <150 x 10^9/L will be administered niraparib 200 mg (2 x 100 mg capsules) daily.
  Other Names: Zejula
Drug: Dostarlimab — Dostarlimab (TSR-042) is administered 500 mg iv Q3W for the first 12 weeks. For the remainder of the study dostarlimab (TSR-042) is administered 1000 mg iv Q6W.
  Other Names: TSR-042

SUMMARY:
This is a multicenter, open-label, non-randomized pilot study (Phase II). The aim is to obtain evidence of efficacy of niraparib and dostarlimab (TSR-042) in patients with relapsed ovarian cancer in two experimental cohorts and to generate data on PARPi (Poly(ADP-ribose)-Polymerase inhibitor) resistance and predictive biomarkers for IO (Immuno-Oncology) and PARPi.

DETAILED DESCRIPTION:
In total, 100 patients are planned to be enrolled in 2 cohorts (60 patients cohort A and 40 patients cohort B).

Cohort A: Recurrent ovarian-, fallopian tube, or primary peritoneal cancer with relapse after more than 6 months of PARPi maintenance therapy.

Cohort B: Recurrent ovarian-, fallopian tube, or primary peritoneal cancer with relapse within 6 months of PARPi maintenance therapy.

All patients must have a known status for BRCA1 and BRCA2 and one or two prior lines of chemotherapy. The last line of chemotherapy should have included platinum.

Both cohorts will receive the selective PARP 1/2 inhibitor niraparib in combination with the anti-PD-1 checkpoint inhibitor dostarlimab (TSR-042) for a maximum treatment duration of 2 years.

The overall objective of this study is to reveal insights in mechanisms of PARPi resistance in epithelial ovarian cancer (EOC) and to obtain preliminary evidence of the efficacy of sequential and/or simultaneous combined immuno-PARPi therapy.

ELIGIBILITY:
Inclusion Criteria:

Cohort A

1. Patients with secondary PARPi resistance, i.e. those whose disease has first relapsed more than 6 months after PARPi maintenance therapy

   a. Criterion for relapse can be according to RECIST 1.1, CA-125 (GCIG) or clinical symptoms

   Cohort B
2. Patients with primary PARPi resistance, i.e. those whose disease has relapsed within 6 months of PARPi maintenance therapy.

   a. Criterion for relapse can be according to RECIST 1.1, CA-125 (GCIG) or clinical symptoms

   Both cohorts
3. Patients with relapsed serous, endometrioid or clear cell epithelial ovarian cancer.
4. Histologically confirmed diagnosis (cytology alone excluded) of high-grade serous, endometrioid or clear cell ovarian carcinoma.
5. Patients with one or two prior lines of chemotherapy. The last line of chemotherapy should have included platinum.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
7. Estimated life expectancy of at least 3 months.
8. Measurable disease according to RECIST or evaluable disease (GCIG CA-125 criteria and other).
9. Urgent chemotherapy not clinically needed according to physicians estimation.
10. Formalin fixed, paraffin-embedded archival tumor available from the primary or recurrent cancer required for all patients.
11. Tumor Biopsy of the relapse is mandatory.
12. Female patients must be >18 years of age.
13. Signed informed consent and ability to comply with treatment and follow-up.
14. Adequate organ function:

    1. Absolute neutrophil count (ANC) ≥1,5 x 10^9/L
    2. Platelets ≥100 x 10^9/L
    3. Hemoglobin ≥9 g/dL
    4. Calculated creatinine clearance ≥60 mL/min using Cockcroft-Gault equation
    5. Total bilirubin ≤1.5 x ULN OR direct bilirubin ≤1 x ULN, patients with documented Gilbert's syndrome total bilirubin ≤2.0 x ULN
    6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN unless liver metastases are present, in which case they must be ≤5 x ULN
15. Adequately controlled blood pressure (BP), with a systolic BP of ≤140 mmHg and diastolic BP of ≤90 mmHg for eligibility. Patients must have a BP of ≤140/90 mmHg taken in the clinic setting by a medical professional within 2 weeks prior to day 1, cycle 1.
16. For women of childbearing potential (WOCBP): agreement to remain abstinent (refrain from heterosexual intercourse) or use a highly effective contraceptive method with a failure rate of <1% per year during the study participation and for at least 6 months after administration of the last dose of medication. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries, fallopian tubes, and/or uterus).

    Examples of contraceptive methods with a failure rate of <1% per year include but are not limited to bilateral tubal ligation and/or occlusion, male sterilization, and intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
17. Negative urine or serum pregnancy test confirmed prior to treatment on day 1.

Exclusion Criteria:

1. Highly symptomatic disease according to physician´s discretion, i.e. rapid remission is required.
2. Patients with mucinous endothelial ovarian cancer.
3. Non-epithelial tumor origin of the ovary, the fallopian tube or the peritoneum (e.g. germ cell tumors).
4. Ovarian tumors of low malignant potential (e.g. borderline tumors).
5. Malignancies other than ovarian cancer (EOC) within 5 years prior to registration, with the exception of those with a negligible risk of metastasis or death (e.g. 5-year OS rate >90%) and treated with expected curative outcome (such as adequately treated non melanoma skin carcinoma, ductal carcinoma in situ, or stage I low grade uterine cancer).
6. More than two prior systemic anticancer regimens; maintenance therapies (e.g. with bevacizumab or PARPi) are not calculated as separate line.
7. More than two lines of PARPi therapies.
8. Administration of other simultaneous chemotherapy drugs, any other anticancer therapy or anti-neoplastic hormonal therapy, or simultaneous radiotherapy during the trial treatment period (hormonal replacement therapy is permitted).

   The following washout requirements for prior therapies/procedures must be observed:

   g. surgery: ≥3 weeks prior to therapy

   h. investigational therapy: within 4 weeks or within less than at least 5 half-lives, whichever is shorter, prior to therapy

   i. radiation: radiation encompassing >20% of bone marrow ≤2 weeks prior to therapy
9. Patient has any known history or current diagnosis of MDS or AML.
10. Prior treatment with immune checkpoint blockade therapies, anti-PD1, or anti-PD-L1 therapeutic antibodies or anti-CTLA4 or anti-TIM-3, or participating in AGO-OVAR 2.29 trial.
11. Treatment with systemic immunostimulatory agents (including but not limited to interferon-alpha (IFN-α) and interleukin-2 (IL-2) within 4 weeks or five half-lives of the drug (whichever is longer) prior to cycle 1, day 1.
12. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 2 weeks prior to cycle 1, day 1, or anticipated requirement for systemic immunosuppressive medications during the trial.

    NOTE: The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g. fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.
13. Administration of a live, attenuated vaccine within 30 days prior to cycle 1, day 1 or anticipation that such a live attenuated vaccine will be required during the study or within 5 months after the last dose of the investigational drugs. Influenza vaccination should be given during influenza season only. Patients must not receive live, attenuated influenza vaccination, for more information see section 5.9.2.
14. Current treatment with anti-viral therapy for HBV.
15. History of idiopathic pulmonary fibrosis (including pneumonitis), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) detected on screening chest CT scan is permitted.
16. Patients with a baseline QT prolongation >470 milliseconds.
17. Patients that are receiving concomitant medications that prolong QTc and are unable to discontinue use for the duration of the study.
18. History or clinical suspicion of brain metastases or spinal cord compression. CT/MRI of the brain is mandatory (within 4 weeks prior to registration) in case of suspected brain metastases. Spinal MRI is mandatory (within 4 weeks prior to registration) in case of suspected spinal cord compression.
19. History of autoimmune disease, including but not limited to dermatomyositis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
20. Immunocompromised patients, e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV). Patients with active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
21. Persistent toxicities (≥CTCAE grade 2) with the exception of alopecia and neurotoxicity CTCAE grade 2.
22. Severe infection requiring oral or IV antibiotics within 4 days prior to registration, including but not limited to active tuberculosis or hospitalization for complications of infection, bacteraemia, or severe pneumonia. Patients receiving prophylactic antibiotics (e.g., to prevent urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
23. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment related complications.
24. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection and posterior reversible encephalopathy syndrome (PRES). This includes also any psychiatric disorder that prohibits obtaining informed consent.
25. Pregnancy, lactation, or intention to become pregnant and Women of childbearing potential (WOBCP) not protected by highly-effective contraceptive methods, including male contraception (e.g. condoms as a barrier method), during the study or within 6 months after the last dose of niraparib or dostarlimab.
26. Known hypersensitivity to infused protein products and to the components of niraparib or dostarlimab.
27. Participant has received colony stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior to initiating protocol therapy.
28. Participant has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted >4 weeks and was related to the most recent treatment.
29. Participant has received a transfusion (platelets or red blood cells) ≤4 weeks prior to initiating protocol therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | At week 16 of treatment
  Defined as Complete Response rate (CR) plus Partial Response Rate (PR) according to RECIST 1.1 assessments

SECONDARY OUTCOMES:
Response Rate | At week 16 of treatment
  Defined as number of patients with Complete Response rate (CR) and Partial Response Rate (PR) according to iRECIST assessments.
Median Progression Free Survival (PFS) | At 6 months
  Defined as the time from randomization to first Progressive Disease (PD) or death, whichever occurs earlier. PD is based on investigators assessment using the Response Evaluation Criteria in Solid Tumors (RECIST 1.1 and iRECIST).
6 months Progression Free Survival (PFS) rate | At 6 months
  Defined as the time from randomization to first progressive disease (PD) or death, whichever occurs earlier. PD is based on investigators assessment using the Response Evaluation Criteria in Solid Tumors (RECIST 1.1 and iRECIST).
Disease Control Rate (DCR) | At 16 weeks
  Defined as sum of Stable Disease (SD), Partial Response (PR) and Complete Response (CR)
Overall Survival (OS) | At 12 months
  Defined as time from start of treatment to death
Time from registration to start of first subsequent therapy (TFST) | Up to approximately 40 months
  Time from registration to start of first subsequent therapy or death, whichever occurs earlier

REFERENCES:
- See also: Homepage of AGO Research GmbH — http://www.ago-ovar.de/